CLINICAL TRIAL: NCT01562197
Title: A Randomized Phase II Clinical Trial on the Efficacy of Axitinib as a Monotherapy or in Combination With Lomustine for the Treatment of Patients With Recurrent Glioblastoma
Acronym: AxiGII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bart Neyns (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Bart Neyns, MD PhD, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AxiGII
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Glioblastoma Multiforme
Keywords: axitinib; glioblastoma; recurrent
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Axitinib; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axitinib (Experimental): axitinib treatment arm
  Interventions: Drug: axitinib
- Axitinib plus Lomustine (Experimental): Axitinib plus Lomustine
  Interventions: Drug: Axitinib plus Lomustine

INTERVENTIONS:
Drug: axitinib — The starting dose of axitinib (AG-013736) is 5 mg BID administered orally with food.
  Other Names: Inlyta (TM)
  Arms: Axitinib
Drug: Axitinib plus Lomustine — Lomustine 90mg/m²
  Other Names: CCNU
  Arms: Axitinib plus Lomustine

SUMMARY:
This clinical trial will recruit patients diagnosed with glioblastoma at the time of recurrence or progression following prior treatment with surgery, radiation therapy and alkylating chemotherapy. Patients will be screened and if found eligible will be randomized to one of two treatment arms (1:1 randomization). Patients randomized to the Axitinib treatment-arm will be treated with Axitinib until progression (they can be treated after progression in the Axitinib plus lomustine arm), unacceptable treatment related toxicity, or patients refusal to continue study treatment. Patients randomized to the Axitinib plus Lomustine-arm will receive treatment until progression, unacceptable treatment related toxicity, or patients refusal to continue study treatment.

ELIGIBILITY:
1. Histopathological diagnosis of glioblastoma (= WHO grade IV glioma of the central nervous system); both "de novo" and "secondary" glioblastoma are eligible;
2. Diagnosis of glioma recurrence or progression following prior treatment with surgery, radiation therapy and alkylating chemotherapy (defined as significant [according to the investigators individual assessment] growth or recurrence of the glioblastoma demonstrated on sequential Gd-MRI before the time of recruitment).
3. The following disease characteristics should be present:

   1. Presence of a measurable tumor lesion that is characterized by gadolinium enhancement on T1-MRI of the brain (with a longest diameter of > 10 mm);
   2. Enhancing characteristics of the glioblastoma as compared to the normal brain on 18F-FET PET (patients with a non-enhancing lesion are not eligible);
   3. No evidence of clinically meaningful spontaneous intra-tumoral hemorrhage on baseline MRI-imaging or in the prior disease history;
4. No contraindication for evaluation by Gd-MRI or 18F-FET PET of the brain;
5. Archival glioma tissue must be available for collection and storage in a centralized tumor bank;
6. An interval of at least 3 months (12 weeks) after the end of prior radiation therapy; and an interval of at least 4 weeks after the last administration of cytotoxic drug treatment (6 weeks in case of administration of a nitrosureum or mitomycin C); and an interval of at least 4 weeks after the last administration of any other kind of anti glioblastoma treatment;
7. A stable dose of corticosteroids for at least 14 days before the initiation of study treatment with axitinib;
8. WHO performance status of 0 or 1;
9. Life expectancy of ≥12 weeks;
10. Male or female, 18 years of age or older;
11. Resolution of all acute toxic effects of prior systemic therapy, radiotherapy or surgical procedure to NCI CTCAEv3.0 grade 0 or 1 or back to baseline except for alopecia or hypothyroidism;
12. Adequate organ function as defined by the following criteria:

    * Total serum bilirubin < 1.5 x ULN (patients with Gilbert's disease exempt)
    * AST and ALT < 2.5 x upper limit of normal (ULN);
    * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥60 mL/min
    * Absolute neutrophil count (ANC) > 1500/mm³ without growth factor support
    * Platelets > 75 000 cells/mm³
    * Hemoglobin ≥9 g/dL (which may be obtained by transfusion or growth factor support)
    * Urinary protein <1+ by urine dipstick. If dipstick is ≥1+ then a 24-hour urine collection should be done and the patient may enter only if urinary protein is <2 grams per 24 hours
13. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.;
14. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception measures during the period of therapy which should be continued for 4 weeks after the last dose of axitinib. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate;
15. No previous treatment on an axitinib trial;
16. No previous treatment with a VEGF or VEGFR-targeted drug (including, but not limited to bevacizumab, aflibercept, cediranib, sorafenib, sunitinib, XL184, and pazopanib);
17. No gastrointestinal abnormalities including:

    1. Inability to take oral medication.
    2. Requirement for intravenous alimentation.
    3. Prior surgical procedures affecting absorption including gastric resection.
    4. Treatment for active peptic ulcer disease in the past 6 months.
    5. Malabsorption syndromes.
    6. Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
18. No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible;
19. No concurrent treatment:

    1. In another therapeutic clinical trial;
    2. With a drug having pro-arrhythmic potential;
    3. With enzyme inducing anti-epileptic drugs (EIAED) within 14 days before dosing with axitinib (e.g. carbamazepine, phenobarbital, phenytoin);
20. No current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine).
21. No current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
22. No requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
23. No active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
24. No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure or any unstable arrhythmia, cerebrovascular accident or transient ischemic attack, within the 12 months prior to study drug administration. No current or recent (within 1 month) use of a thrombolytic agent or a thrombo-embolic event;
25. No known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness;
26. No serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment;
27. No history of a malignancy (other than glioma) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years;
28. No major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks of treatment. (Also excluded are patient with fine needle aspirations within 7 days of treatment);
29. No pregnancy or breastfeeding;
30. No history of hemoptysis > ½ tsp of bright red blood per day within past 1 week;
31. No other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
32. No dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol;
33. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment;
34. Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other study procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-04; Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
anti-tumor effect of axitinib as a single therapeutic agent and in combination with Lomustine | 6months
  To estimate the anti-tumor effect of axitinib as a single therapeutic agent for the treatment of glioblastoma patients at the time of recurrence/progression following prior surgery, radiation and alkylating chemotherapy and in combination with Lomustine

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium